CLINICAL TRIAL: NCT06815978
Title: Validation of ESPEN-EASO Algorithm for the Diagnosis of Sarcopenic Obesity (SO)
Brief Title: Validation of an Algorithm for the Diagnosis of Sarcopenic Obesity
Status: Recruiting | Type: Observational
Sponsor: Elisa Giannetta (Other)
Collaborators: ministero della ricerca e dell'università (Unknown)
Responsible Party: Sponsor-Investigator, Elisa Giannetta, Associate Professor, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: PRIN-202229ET3S
Record Dates: First submitted 2024-11-07; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenic Obesity
Keywords: Sarcopenic obesity; obesity; nutrition; gut microbiome; diagnostic ciriteria
MeSH Terms: conditions — Obesity | interventions — Ultrasonography; Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — * faeces
  * blood samples
  * urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient with sarcopenic obesity
  Interventions: Diagnostic Test: DXA; Diagnostic Test: ultrasonography; Diagnostic Test: indirect calorimetry; Diagnostic Test: MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy); Diagnostic Test: bioimpedentiometry
- Patients with obesity
  Interventions: Diagnostic Test: DXA; Diagnostic Test: ultrasonography; Diagnostic Test: indirect calorimetry; Diagnostic Test: MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy); Diagnostic Test: bioimpedentiometry

INTERVENTIONS:
Diagnostic Test: DXA — Dual energy X-ray absorptiometry
Diagnostic Test: ultrasonography — ultrasonography
Diagnostic Test: indirect calorimetry — indirect calorimetry
Diagnostic Test: MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy) — MRI/ MRS (Magnetic Resonance Imaging /Magnetic Resonance Spectroscopy)
Diagnostic Test: bioimpedentiometry — bioimpedentiometry

SUMMARY:
The proposed research project aims to investigate sarcopenic obesity (SO), a condition characterized by the combination of high body fat and low skeletal muscle mass, with a focus on muscle function. SO has been defined according to the ESPEN-EASO algorithm, and this study aims to evaluate its validity, exploring associations with circulating biomarkers and functional outcomes. By enrolling 75 subjects with SO and a control sample of 75 subjects with non-sarcopenic obesity, the primary objective of this study is to examine the consistency of the proposed diagnostic criteria with respect to circulating biomarkers and functional outcomes. Secondary objectives include the assessment of additional variables and the detailed profiling of SO subjects through questionnaires and multidimensional tests. The ethical aspect of the present study will be guaranteed through written informed consent and protection of privacy, respecting international regulatory standards. The investigators believe that this work provides significant contributions to the understanding of sarcopenic obesity and to the validation of diagnostic criteria, with possible implications for public health. The investigators are available for further clarifications and approvals required by the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* BMI equal more than 30
* Caucasians

Exclusion Criteria:

* any disease or medication that can significantly affect body composition (eg.malignant diseases in the last 5 years, autoimmune diseases, neurological diseases, syndromic obesity),
* level of physical activity more than 3 METS
* alcohol intake more than 140g/wk for M and 70g/wk for F
* participation in a weight-reducing program (last 3 months),
* impossibility to perform DXA exam
* pregnancy and breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical setting from Azienda Policlinico Umberto I, Rome, Italy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Association between diagnostic criteria for Sarcopenic Obesity and hemochrome in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and ferritin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and transferrin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and iron in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and AST in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and ALT in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and GGT in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and alkaline phosphatase in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and total bilirubin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and fractionated bilirubin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and triglyceride in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and free fatty acid (FFA) in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and total cholesterol in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and HDL-Cholesterol in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and LDL-Cholesterol in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Apo A1 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Apo B in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and serum creatinine in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and blood urea nitrogen in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and total proteins in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and albumin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and pseudocholinesterase in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and vitamin D3 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Vitamin B12 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Vitamin B6 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Hs-CRP in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Atrial Natriuretic Peptide (ANP) in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Brain Natriuretic Peptide in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and standard OGTT glycaemia in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and standard OGTT insulin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and C-peptide in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and TSH in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and FT3 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and FT4 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and GH in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and IGF-1 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and acylated ghrelin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and unacylated ghrelin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and testosterone (in men) in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and estradiol (in women) in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and adrenal-derived dehydroepiandrosterone in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and myostatin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and leptin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and adiponectin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Irisin in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and parathormone in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and cortisol in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and sodium in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and potassium in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and calcium in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and phosphorus in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and chloride in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and magnesium in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and TNF-α in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and interleukine 6 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and interleukine 8 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and interleukine 10 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and interleukine 15 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and interleukine 18 in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and hand-grip strength test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and 5- time sit-to-stand test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and balance test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Gait speed 4m in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and 6-minute walk test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Knee extension strenght in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Sit and reach test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Time up and go test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and One-Leg Standing balance in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and 30s chair stand test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and Joint mobility test in Odd Ratios as assessed by Multivariate analysis | baseline, 6 month

SECONDARY OUTCOMES:
Association between diagnostic criteria for Sarcopenic Obesity and Energy expenditure in Odd Ratios as assessed by multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and body fat percentage (assessed by DXA) in Odd Ratios as assessed by multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and body fat percentage (assessed by BIA) in Odd Ratios as assessed by multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and skeletal muscle mass (assessed by BIA) in Odd Ratios as assessed by multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and appendicular lean mass to weight in Odd Ratios as assessed by multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and bone mineral density in Odd Ratios as assessed by multivariate analysis | baseline, 6 month
Association between diagnostic criteria for Sarcopenic Obesity and visceral adipose tissue (assessed by DXA) in Odd Ratios as assessed by multivariate analysis | baseline, 6 month

OTHER OUTCOMES:
weight in Kilograms | on enrollment day and at the end of the intervention (6 month)
Height in meters | on enrollment day and at the end of the intervention (6 month)
calf circumference in centimeters | on enrollment day and at the end of the intervention (6 month)
mid-arm muscle circumference in centimeters | on enrollment day and at the end of the intervention (6 month)
waist circumference in centimeters | on enrollment day and at the end of the intervention (6 month)
Risk of Sarcopenia as assessed by SARC-F Questionnaire | on enrollment day and at the end of the intervention (6 month)
hand-grip strength in kilograms as assessed by Jamar Dynamometer mod.5030J1 | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in seconds as assessed by 5 time sit-to-stand test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in seconds as assessed by balance test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in seconds as assessed by 4m-Gait speed test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in meters as assessed by 6-minute walk test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in kilograms as assessed by Knee extension strength test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in seconds as assessed by Sit and reach test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in seconds as assessed by Time up and go test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in seconds as assessed by One-Leg Standing balance test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in repetitions as assessed by 30s chair stand test | on enrollment day and at the end of the intervention (6 month)
lower limb functionality in radiants as assessed by Joint mobility test. | on enrollment day and at the end of the intervention (6 month)
body fat percentage in percentage as assessed by DXA | on enrollment day and at the end of the intervention (6 month)
body fat percentage in percentage as assessed by BIA | on enrollment day and at the end of the intervention (6 month)
skeletal muscle mass in kilograms as assessed by BIA | on enrollment day and at the end of the intervention (6 month)
appendicular lean mass to weight in kilograms/kilograms as assessed by DXA | on enrollment day and at the end of the intervention (6 month)
bone mineral density in Z-score as assessed by DXA | on enrollment day and at the end of the intervention (6 month)
visceral adipose tissue in grams as assessed by DXA | on enrollment day and at the end of the intervention (6 month)
epicardial fat in millimeters as assessed by Transthoracic echocardiogram | on enrollment day and at the end of the intervention (6 month)
left ventricular mass in grams as assessed by Transthoracic echocardiogram | on enrollment day and at the end of the intervention (6 month)
carotid Intima-Media thickness in millimeters as assessed by Carotid ultrasonography | on enrollment day and at the end of the intervention (6 month)
fat inltration in percentage as assessed by MRI | on enrollment day and at the end of the intervention (6 month)
Energy expenditure in Kilocalories as assessed by Cosmed Q-NRG | on enrollment day and at the end of the intervention (6 month)
Energy expenditure in METs as assessed by Actigraph GT9X | on enrollment day and at the end of the intervention (6 month)
proton density fat fraction in percentages assessed by magnetic resonance imaging | on enrollment day and at the end of the intervention (6 month)
Energy expenditure in METs/min/week as assessed by IPAQ Questionnaire | on enrollment day and at the end of the intervention (6 month)
Visual Analog Score for disability level as assessed by TSD-OC Questionnaire | on enrollment day and at the end of the intervention (6 month)
Quality of Sleep in a 24-point scale as assessed by The Epworth Sleepiness Scale | on enrollment day and at the end of the intervention (6 month)
Adherence to Mediterranean Diet in a 218-point scale as assessed by DISC-MED Questionnaire | on enrollment day and at the end of the intervention (6 month)
Nutrition Knowledge in a 88-point scale as assessed by I-NK Questionnaire | on enrollment day and at the end of the intervention (6 month)
Socio Economic Factors in 220-point scale assessed by SEF Questionnaire | on enrollment day and at the end of the intervention (6 month)
Hemochrome in g/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Ferritin in µg/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Transferrin in g/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Iron in µmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
AST in U/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
ALT in U/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
GGT in U/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
alkaline phosphatase in U/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
total bilirubin in mg/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
fractionated bilirubin in mg/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Triglycerides in mmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Free Fat Acids (FFA) in mmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Total cholesterol in mmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
HDL-cholesterol in mmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
LDL-cholesterol in mmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Apo A1 in g/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Apo B in g/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Serum creatinine in mg/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Blood urea nitrogen in mmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Total proteins in g/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Albumin in g/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Pseudocholinesterase in U/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Vitamins: D3 in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Vitamin B12 in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Vitamin B6 in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Hs-CRP in mg/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
BNP in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
ANP in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Standard OGTT (glycaemia) in mmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Standard OGTT (insulin) in pmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
C-peptide in pmol/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
TSH in µU/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
FT3 in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
FT4 in ng/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
GH in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
IGF-1 (Insulin-like Growth Factor 1) in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Ghrelin in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
testosterone (in men) in ng/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Estradiol (in women) in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
dehydroepiandrosterone (DHEA) in µg/dLassessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
myostatin in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
leptin in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
adiponectin in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
irisin in ng/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
parathyroid hormone (PTH) in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
cortisol in µg/dL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
sodium in mEq/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
potassium in mEq/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
calcium in mEq/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
chloride in mEq/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Phosphorus in mEq/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Magnesium in mEq/L assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
TNF-α (Tumor Necrosis Factor-alpha) in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Interleukin 6 in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Interleukin 8 in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Interleukin 10 in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Interleukin 15 in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)
Interleukin 18 in pg/mL assessed by human blood biochemistry analyzer | on enrollment day and at the end of the intervention (6 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Policlinico Umberto I, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No